CLINICAL TRIAL: NCT04148040
Title: Per-oral Pyloromyotomy for Treating Infantile Hypertrophic Pyloric Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSLQL
Record Dates: First submitted 2019-10-12; First posted 2019-11-01 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Infantile Hypertrophic Pyloric Stenosis; Pyloromyotomy
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic | interventions — Pyloromyotomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- G-POEM for infantile hypertrophic pyloric stenosis (Experimental): The procedure includes four steps: a) a transversal mucosal incision was performed at the proximal antrum. b) a submucosal longitudinal tunnel was created across the pyloric ring. c) full-thickness pyloromyotomy was performed, with a little extension of the antrum. After pyloromyotomy, an ultrathin gastroscope was used to inspect the mucosa and pyloric outlet. d) after careful hemostasis, the mucosal entry was closed by clips.
  Interventions: Procedure: G-POEM

INTERVENTIONS:
Procedure: G-POEM — Per-oral pyloromyotomy (POP), also named as gastric per-oral endoscopic myotomy (G-POEM), for treating infantile hypertrophic pyloric stenosis (IHPS) has the following steps: mucosal incision, creation of submucosal tunnel, full-thickness pyloromyotomy, closure of the mucosal entry.

SUMMARY:
Infantile hypertrophic pyloric stenosis (IHPS) is the most common condition for surgical treatment in infant. Traditionally, laparoscopic or open pyloromyotomy are the standard treatments. However, because of severe dehydration, electrolyte disturbance, and malnutrition, these patients have lower tolerance about surgery and recover more slowly than usual. We are going to study the per-oral pyloromyotomy (POP), also named as gastric per-oral endoscopic myotomy (G-POEM), which showed promising results for adult gastroparesis, for a novel application of treating IHPS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pyloric stenosis with or without sonographic confirmation.

Exclusion Criteria:

* Comorbid conditions that could affect postoperative recovery.
* Needed an additional procedure during the same anaesthetic.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
episodes of postoperative vomiting | 6 months after surgery
  Primary outcomes included episodes of postoperative vomiting in times.
major complication | 6 months after surgery
  Primary outcomes included major complication in times (based on lexicon and Clavien-Dindo classification, eg, vital-sign instability, ICU stay, hospital readmission, conversion to laparoscopic or open pyloromyotomy, invasive postoperative procedure, haemorrhage, blood transfusion, or prolonged hospitalization due to functional impairment).

SECONDARY OUTCOMES:
operating and anaesthetic time | 6 months after surgery
  Secondary outcomes included operating and anaesthetic time in minutes.
myotomy length | 6 months after surgery
  Secondary outcomes included myotomy length in centimeters
other complications | 6 months after surgery
  Secondary outcomes included other complications (yes or no) (eg, mucosal injury, delayed mucosal barrier failure, incomplete pyloromyotomy, and respiratory complications without invasive intervention).
postoperative pain assessment by "Pain assessment for children under four years" | 6 months after surgery
  Secondary outcomes included postoperative pain assessment in score.
  This measurement chart is "Pain assessment for children under four years" which of pain scoring in the postoperative set up is:
  Cry (yes or no), Posture (relaxed or tense), Expression (relaxed, happy or distressed), Response when spoken to (yes or no).
  (Gupta A, Kaur K, Sharma S, Goyal S, Arora S, Murthy RS. Clinical aspects of acute post-operative pain management & its assessment. J Adv Pharm Technol Res. 2010;1(2):97-108.)
analgesia requirements | 6 months after surgery
  Secondary outcomes included analgesia requirements (yes or no).
time to full enteral feed | 6 months after surgery
  Secondary outcomes included time to full enteral feed in hours.
postoperative length of stay | 6 months after surgery
  Secondary outcomes included postoperative length of stay in days.
need for re-operation | 6 months after surgery
  Secondary outcomes included need for re-operation (yes or no).

CONTACTS AND LOCATIONS:
Overall Officials: Pinghong Zhou, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan hospital, Shanghai, China